CLINICAL TRIAL: NCT02073396
Title: Assessment of Thrombotic Status in Patients at Risk of Cardiovascular Thrombosis
Status: Completed | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof Diana Gorog, MD, PhD, FRCP, East and North Hertfordshire NHS Trust
Other Study IDs: No 1.1; 4 Dec 2012; REC 12/EE/0466 (Other: NRES Committee East of England - Essex, UK)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: Patients diagnosed with coronary disease or atrial fibrillation. All the patients will undergo Global Thrombosis Test.
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Patients will undergo the tests of thrombosis, before and after stabilisation of their cardiac condition. Cardiac stabilisation will be provided by clinical cardiac teams, outside and independently from the study.

SUMMARY:
Patients with coronary artery disease (CAD) and atrial fibrillation (AF) are at increased risk of stroke and heart attack. Such events are usually caused by increased stickiness of the blood causing a blood clot to block the artery (thrombus) in the heart or the brain. The aim of this study is to assess the stickiness of the blood (global thrombotic status) in patients with CAD and AF at baseline and after clinical stabilisation to see how disease state and clinical treatments affect the stickiness of the blood (thrombotic status). This will be a single centre study. Patients diagnosed with CAD or AF will have a blood sample taken at baseline and after clinical stabilisation. Blood stickiness will be tested with the Global Thrombosis Test. The results will be evaluated to assess the effect of disease process and clinical state on blood stickiness to gain further understanding of this condition and form the basis for future studies aimed at identifying patients who are at high risk of future cardiovascular events, based on increased blood stickiness.

DETAILED DESCRIPTION:
Impaired thrombotic status is associated with adverse cardiovascular events. Patients with coronary artery disease (CAD) and atrial fibrillation (AF) are at increased risk of thrombotic events. It is not known whether thrombotic status differs in these patients, or how thrombotic status alters in response to clinical stabilisation with treatment.

The aim of this study is to assess the global thrombotic status (stickiness of the blood) in patients with coronary artery disease and atrial fibrillation at baseline and after clinical stabilisation.

This is a small, pilot, hypothesis-generating study. Design Single centre, hypothesis-generating study. Patients diagnosed with coronary disease (n=70) or atrial fibrillation (n=70) recruited from amongst in-patients or out-patients, will have a blood draw at presentation and after clinical stabilisation. Blood will be tested to assess global thrombotic status.

The recruitment period is 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 years or over.
2. Patients diagnosed with CAD or AF and free of exclusion criteria below.
3. Not actively using tobacco products (due to vasoactive and pro-aggregatory effects of nicotine).
4. The participant is willing and able to understand the Subject Information Sheet and provide informed consent.
5. The participant must agree to comply with the drawing of blood samples for the assessments.

Exclusion Criteria:

1. Male and female participants aged < 18 years of age.
2. Patients with impaired renal function eGFR <30 ml/min (since renal failure is associated with platelet function defect that may confound results).
3. The participant has, in the opinion of the investigator, significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, haemorrhagic metabolic or other disease likely to confound the study requirements or analyses.
4. The participant has a gives a history of substance abuse or demonstrates signs or clinical features of active substance abuse or psychiatric disease.
5. Alcohol consumption above recommended safe levels (i.e. more than 21 units per week for males, or more than 14 units per week for females) due to the potential effects of high alcohol levels on platelet reactivity.
6. Any illness deemed significant by the investigator during the four (4) weeks preceding the screening period of the study.
7. Any major bleeding diathesis or blood dyscrasia (platelets < 70 x 109/l, Hb <8 g/dl, INR>1.4, APTT> x 2UNL, leucocyte count< 3.5x 109/l, neutrophil count < 1x 109/l)
8. Currently enrolled in an investigational device or drug trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with coronary disease or atrial fibrillation. Participants will be recruited from amongst in-patients or out-patients
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The occlusion and lysis time. | 1-3 months
  The occlusion and lysis timet.

SECONDARY OUTCOMES:
no secondary outcome measures to be identified | no secondary outcome measures to be identified
  no secondary outcome measures to be identified

OTHER OUTCOMES:
no other outcome measures to be identified | no other outcome measures to be identified
  no other outcome measures to be identified

CONTACTS AND LOCATIONS:
Overall Officials: Diana A Gorog, Prof, Principal Investigator — East & North Herts NHS Trust
Locations (1):
- East & North Herts NHS Trust (Queen Elizabeth II Hospital, Howlands, Welwyn Garden City, AL7 4HQ and Lister Hospital, Coreys Mill Lane, Stevenage, Herts , SG1 4AB -those two hospitals operate as one institution, Stevenage, Herts, United Kingdom